CLINICAL TRIAL: NCT01900860
Title: Randomized Double-blind Study Investigating Dose-dependent Longitudinal Effects of Vitamin D Supplementation on Bone Health
Brief Title: Dose-dependent Effects of Vitamin D on Bone Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Pure North S'Energy Foundation (Other)
Responsible Party: Principal Investigator, David A. Hanley, MD, FRCPC, Professor Emeritus, Department of Medicine, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20130101
Record Dates: First submitted 2013-07-02; First posted 2013-07-17 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Age-Related Osteoporosis
Keywords: Vitamin D; Bone quality; Bone density; calcium metabolism; High resolution peripheral quantitative computed tomography; Dual X-ray absorptiometry; Quality of life
MeSH Terms: conditions — Osteoporosis | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- vitamin D 10,000 IU (Active Comparator): Subjects in this arm receive 10,000 IU Vitamin D p.o. (as 5 drops of a blinded vitamin D solution) per day. Duration: 3 years
  Interventions: Dietary Supplement: Vitamin D
- Vitamin D 4000 IU (Active Comparator): Subjects in this arm receive 4,000 IU Vitamin D p.o. (as 5 drops of a blinded vitamin D solution) per day. Duration: 3 years
  Interventions: Dietary Supplement: Vitamin D
- Vitamin D 400 IU (Active Comparator): Subjects in this arm receive 400 IU Vitamin D p.o. (as 5 drops of a blinded vitamin D solution) per day. Duration: 3 years
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Three different doses of vitamin D will be administered in a double-blinded fashion. The three doses are 400, 4000, or 10,000 IU/day
  Other Names: Vitamin D3, Cholecalciferol

SUMMARY:
We propose to conduct a randomized double blind trial of three doses of vitamin D, 400, 4000, and 10,000 International Units (IU) per day, to assess the effect on bone density and architecture as assessed by high resolution peripheral quantitative tomography (HR-pQCT) measurements at the radius and distal tibia, and standard Dual X-ray absorptiometry (DXA). Other measures of bone and calcium metabolism will be assessed. The trial will last as long as three years. Approximately 300 healthy men and women, aged 50-70 years of age, will be recruited, and randomly assigned to one of the three doses of vitamin D. Other outcome variables assessed include quality of life, depression, muscle strength and balance.

DETAILED DESCRIPTION:
Hypotheses being tested:

1. It is hypothesized that vitamin D, in a dose-dependent manner, will suppress parathyroid hormone action, resulting in less bone turnover, and decreased cortical porosity, leading to improved bone strength as assessed by finite element analysis.
2. It is hypothesized that vitamin D, in a dose-dependent manner, will increase bone density in the central skeleton (spine, hip), as measured by the current standard method of dual X-ray absorptiometry (DXA).
3. It is hypothesized that vitamin D, in a dose-dependent manner, will have an impact on quality of life, including indices of depression, as measured by the SF-36 questionnaire and an appropriate index of depression.

Outcomes:

Primary outcomes:

* (1) bone density and (2) strength as measured by HR-pQCT

Secondary outcomes:

* HR-pQCT assessment of bone microarchitecture, examining the relative contribution of trabecular and cortical bone. We have chosen four parameters for statistical analysis, and have listed them as secondary outcome variables in the section below: cortical density, cortical porosity, trabecular density and trabecular number.
* bone mineral density as measured by DXA
* parameters of calcium metabolism, including biochemical markers of bone turnover and DNA to examine possible variations in the genes that control vitamin D metabolism.
* quality of life score
* depression scale score
* balance, grip strength.
* fasting glucose and Hemoglobin A1C will also be measured.
* Safety will be assessed during the scheduled follow-up visits by obtaining history of adverse events, as well as measurements of serum and urine parameters of mineral metabolism as described below.

INTERVENTION DRUG: Vitamin D3 in one of three doses Rationale: For adults under age 70 years, the recent Institute of Medicine (IOM) report recommends a total intake of 600 IU vitamin D/day will provide all the vitamin D needed for bone health, and since the typical Canadian diet contains between 200 and 300 units of vitamin D, the subjects in the lowest dose arm of our study will receive 400 IU/day. The other two groups will receive 10,000 IU and 4,000 IU, respectively. The 10,000 IU dose is the tolerable upper intake level (TUL) recommended by Hathcock et al (Am J Clin Nutr 2007) and 4,000 IU is the IOM's recommended TUL.

Calcium intake:

All subjects will have adequate calcium intake as defined by the Institute of Medicine (total of 1200 mg/day). A brief dietary history will be taken and subjects will be instructed to take an appropriate dose of supplemental calcium if their daily intake is less than 1200 mg/day (the IOM's Recommended Daily Allowance for this study population).

Interim analysis (with maintenance of blinding of subjects and investigators as to treatment arm):

* planned at and of years 1 and 2, as well as the final analysis at year 3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women and men between 55 and 70 years of age; women will be at least 5 years post-menopause. Presence of a chronic illness does not exclude participation if the condition is stable and managed by a physician.
* Baseline lumbar spine and total hip bone mineral density (BMD) T-score above 2.5 as assessed using dual x-ray absorptiometry (DXA).

Exclusion Criteria:

* A serum 25-[OH] vitamin D (25OHD) of <30 nmol/L (<12 ng/mL) or >125 nmol/L (50 ng/mL).
* Hypercalcemia (serum calcium >2.55 mmol/L), hypocalcemia (serum calcium <2.10 mmol/L) or eGFR <30 mL/min.
* Surgical cure of Primary Hyperparathyroidism within the last year.
* Active kidney stone disease (recurrent stones, recent kidney stone [within last 2 years])
* Known hypersensitivity or allergy to Vitamin D
* Serum creatinine, AST, ALT, PTH, calcium, or alkaline phosphatase greater than 1.5 times the upper limit of normal at the screening visit
* BMD exclusions:

  1. High 10-year risk for osteoporotic fracture, as defined by the Canadian Association of Radiologists/Osteoporosis Canada calculator, or the World Health Organization's FRAX calculator.
  2. DXA T-score below or equal to -2.5 SD.
* Have taken bone active osteoporosis prescription drugs in the past 2 years (bisphosphonates) or 1 year (other osteoporosis prescription therapies).
* Any medical condition that would prevent participation in a clinical trial for a full three years.
* Medications such as prednisone >2.5 mg daily (or equivalent); other bone active medications such as tamoxifen or aromatase inhibitors for breast cancer, or androgen deprivation therapy of prostate cancer.
* Disorders known to affect vitamin D metabolism such as sarcoidosis or renal failure or malabsorption disorders (e.g. pancreatic insufficiency or celiac disease).
* Regular (monthly or more frequent) use of tanning salons.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2013-08; Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Total Bone Mineral Density (Tt.BMD) at the distal radius and tibia, as measured by High Resolution peripheral Quantitative Tomography (HR-pQCT) | Participants will be followed from baseline up to 36 months
  Unlike the measurement of bone density by DXA (a secondary outcome, see below), which estimates bone density based on assumptions of the depth of a 2-dimensional image of bone, HR-pQCT measurement of Tt.BMD provides a true volume based density measurement. HR-pQCT also provides a much higher resolution image of the region of interest than the image derived from a DXA measurement.
  Units of this measurement are milligrams hydroxyapatite per cubic centimetre (mg HA/cm3).
  The analysis will examine change in Tt.BMD at distal radius and tibia from baseline to measurements at 6, 12, 24, and 36 months.
Bone strength, as estimated by Finite Element Analysis of High Resolution peripheral Quantitative Computed Tomography (HR-pQCT) measurements at the distal radius and tibia | Participants will be followed from baseline up to 36 months
  HR-pQCT scans provide the ability to measure a true volumetric density of the bone region of interest and to study microarchitecture of both trabecular and cortical bone, from which an assessment of strength by Finite Element Analysis (FEA) can be determined: briefly, a 3-dimensional computer model of bone can be constructed from the HR-pQCT data, and subjected to strength testing. FEA software (FAIM, version 6.0, Numerics88 Solutions, Calgary, Canada) is used to estimate failure load (N) based on 2 % of the elements exceeding 7,000 μstrain.
  The analysis examines change from baseline measured at 6, 12, 24, and 36 months.

SECONDARY OUTCOMES:
Cortical bone density (Ct.BMD) of bone as measured by HR-pQCT | From baseline to 36 months - measured at 0, 6, 12, 24, and 36 months.
  Cortical density (Ct.BMD) is a morphological parameter of microarchitecture of bone, and is measured in mg HA/cm3
Cortical Porosity (Ct.Po) of bone as measured by HR-pQCT | From baseline to 36 months - measured at 0, 6, 12, 24, and 36 months.
  Cortical Porosityis a morphological parameter of microarchitecture of bone, and is measured in percent.
Trabecular bone density (Tb.BMD) of bone as measured by HR-pQCT | From baseline to 36 months - measured at 0, 6, 12, 24, and 36 months.
  Trabecular density (Tb.BMD) is a morphological parameter of microarchitecture of bone, and is measured in mg HA/cm3
  Trabecular density (Tb.BMD) is a morphological parameter of microarchitecture of bone, and is measured in mg HA/cm3
Trabecular number (Tb.N) as measured by HR-pQCT | From baseline to 36 months - measured at 0, 6, 12, 24, and 36 months.
  Trabecular number (Tb.N) is a morphological parameter of microarchitecture of bone, and is measured as mean number of trabeculae per unit of length (mm)
Bone Mineral Density as measured by Dual X-ray Absorptiometry | Participants will be followed from baseline up to 36 months
  Dual X-ray absorptiometry (DXA) will be used to scan the distal radius, lumbar spine and the proximal femur to obtain an areal (two dimensional) estimate of bone mineral density (aBMD). DXA is the current clinical standard for measuring bone density. From the scan of the lumbar spine and left proximal femur (~ 1 min), aBMD (g/cm2) will be used to determine a subject-specific T-score (aBMD compared to reference mean for a young healthy adult) and this value will be compared to standard World Health Organization criteria to classify each subject as normal (T-score>-1), low bone density (-1 < T > -2.5) or osteoporotic (T score < -2.5). Change from baseline will be assessed at 12, 24 and 36 months.
Quality of Life (Mental Health Component) | Participants will be followed from baseline up to 36 months
  Vitamin D deficiency has been associated with depression. We propose to examine whether our Vitamin D intervention has an effect on depression or other aspects of mental health. The SF-36 questionnaire will be administered at baseline and at 12, 24, and 36 months. This will be used to assess subjects' perception of their Quality of Life, specifically the Mental Health Component, and whether the intervention (Vitamin D dose assignment) is associated with changes in the SF-36 scores for Mental Health Component change over the course of the study.
Depression symptoms | Participants will be followed from baseline up to 36 months
  PHQ-9 questionnaire will be used to assess any effect the Vitamin D intervention might have on depression symptoms. The PHQ-9 analog scale score will be measured at entry and at 3, 6 and 12 months, then annually. This is not expected to be a safety issue in recruiting healthy volunteers, but obviously could become one.
Biochemical markers of calcium and bone metabolism | Participants will be followed from baseline up to 36 months
  In addition to the markers identified as safety measures in "other outcomes" (serum and urine calcium, serum creatinine, etc), we will also obtain serum for measurement of markers of bone turnover: serum C-telopeptide of Type I Collagen (CTX), and Procollagen I N-terminal Propeptide. Measurements taken at baseline and at 3, 6, 12, 24, and 36 months. Still to be arranged: Under-carboxylated osteocalcin and osteocalcin.
Balance and grip strength | Participants will be followed from baseline up to 36 months
  The balance tests include standing with (a) two feet on the force platform with eyes open, (b) two feet on the force platform with eyes closed, (c) two feet on a foam pad with eyes open, and (d) two feet on a foam pad with eyes closed. All tests will be performed 3 times, and a blindfold will be used for all eyes-closed assessments. The total testing time is approximately 15 minutes. Measurements done at baseline and at 12, 24 and 36 months

OTHER OUTCOMES:
Safety: changes in parameters of calcium metabolism | Participants will be followed from baseline up to 36 months
  The main concern in safety of vitamin D consumption is the avoidance of toxicity in the form of hypercalcemia or renal damage, related to hypercalcemia and hypercalciuria. Two of the doses in this study are generally accepted as safe. The 10,000 IU daily dose exceeds the recommended upper limit of safe, unsupervised vitamin D intake, hence, this trial includes regular clinical laboratory testing of parameters of calcium metabolism, including serum and urine calcium, parathyroid hormone, 25OH-Vitamin D. Measurements will be done at baseline, 3, 6, 12, 24, and 36 months
Safety: Parameters of glucose metabolism | Participants will be followed from baseline up to 36 months
  Hemoglobin A1C, and fasting glucose, and the osteocalcin measurements will address some of the potential effects of vitamin D on glucose metabolism. A full assessment of the effects of vitamin D on diabetes and glucose metabolism is beyond the scope of this proposal, but because these parameters are very easily obtained measurements they will be examined at baseline, 3, 6 , 12, 24 and 36 months.
Safety: Peripheral Vascular Calcification, as assessed by HR-pQCT at the distal radius and tibia | Participants imaging studies will be followed from baseline up to 36 months
  Recently, it has become apparent that the HRpQCT images obtained at the distal radius and tibia include enough detail of the arteries providing blood supply to the hand and foot, that quantification of calcification of the medial layer of these blood vessels (radial and ulnar arteries, anterior and posterior tibial arteries), may be possible. Vitamin D might play a role in vascular calcification (animal models suggest protection; vitamin D toxicity may be associated with soft tissue calcification). Consequently, the range and duration of vitamin D Dose in this protocol may allow discovery of a vitamin D effect on calcium deposition.
  Reference: Patsch JM, Zulliger MA, Vilayphou N, et al. Quantification of lower leg arterial calcifications by high-resolution peripheral quantitative computed tomography. Bone. 2014 Jan;58:42-7.

CONTACTS AND LOCATIONS:
Overall Officials: David A Hanley, MD, FRCPC, Principal Investigator — The University of Calgary; Steven K Boyd, PhD, Principal Investigator — The University of Calgary
Locations (1):
- The University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burt LA, Gaudet S, Kan M, Rose MS, Billington EO, Boyd SK, Hanley DA. Methods and procedures for: A randomized double-blind study investigating dose-dependent longitudinal effects of vitamin D supplementation on bone health. Contemp Clin Trials. 2018 Apr;67:68-73. doi: 10.1016/j.cct.2018.02.009. Epub 2018 Feb 20. PMID 29471124
- [Derived] Burt LA, Billington EO, Rose MS, Kremer R, Hanley DA, Boyd SK. Adverse Effects of High-Dose Vitamin D Supplementation on Volumetric Bone Density Are Greater in Females than Males. J Bone Miner Res. 2020 Dec;35(12):2404-2414. doi: 10.1002/jbmr.4152. Epub 2020 Sep 16. PMID 32777104
- [Derived] Billington EO, Burt LA, Plett R, Rose MS, Boyd SK, Hanley DA. Effect of high-dose vitamin D supplementation on peripheral arterial calcification: secondary analysis of a randomized controlled trial. Osteoporos Int. 2020 Nov;31(11):2141-2150. doi: 10.1007/s00198-020-05500-2. Epub 2020 Jun 15. PMID 32556518
- [Derived] Billington EO, Burt LA, Rose MS, Davison EM, Gaudet S, Kan M, Boyd SK, Hanley DA. Safety of High-Dose Vitamin D Supplementation: Secondary Analysis of a Randomized Controlled Trial. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgz212. doi: 10.1210/clinem/dgz212. PMID 31746327
- [Derived] Burt LA, Billington EO, Rose MS, Raymond DA, Hanley DA, Boyd SK. Effect of High-Dose Vitamin D Supplementation on Volumetric Bone Density and Bone Strength: A Randomized Clinical Trial. JAMA. 2019 Aug 27;322(8):736-745. doi: 10.1001/jama.2019.11889. PMID 31454046